CLINICAL TRIAL: NCT05545982
Title: Comparison of Video Laryngoscope Using Miller or Macintosh Approach During Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Han-Liang Chiang, Director of Cardiothoracic Anesthesiology, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS19-CT9-11
Record Dates: First submitted 2022-09-07; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Difficult Intubation
Keywords: difficult intubation; video laryngoscope

STUDY DESIGN:
Intervention Model Description: one-group pretest-posttest study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intubation with Miller approach (Experimental): Posttest group: Patient receive intubation with conventional video laryngoscope with Miller approach.
  Pretest group: Patient receive intubation with conventional video laryngoscope with Macintosh approach.
  Interventions: Procedure: Video laryngoscope with Miller approach

INTERVENTIONS:
Procedure: Video laryngoscope with Miller approach — Miller approach indicates lifting epiglottis during laryngoscopy, which is the way of using Miller laryngoscope

SUMMARY:
Video laryngoscope has become recommended option during difficult intubation. Guidelines of ASA at 2013 had suggested using video laryngoscope after failure intubation of direct laryngoscope. Varieties of video laryngoscope had been invented with different curves. We call the one which has the same curve of Macintosh laryngoscope as conventional video laryngoscope in this study. Mostly, the way of using conventional video laryngoscope is suggested as Macintosh method. However, with the front positioning camera, Miller method can theoretically improve the glottic opening. We intend to discuss whether using Miller approach with conventional video laryngoscope can improve glottic opening or not.

DETAILED DESCRIPTION:
Video scope can provide better glottic opening by increase the tilting angle of the tip, and the position of camera can provide larger vision angle. However, while the angle increases, the endotracheal tube must fallow the curve, which may require learning curve of the operator. In Glidescope as example, increase the tilting angle can help with glottic exposure, however the steep curve will simultaneously increase the difficulty of inserting the tube or using Magill forceps, especially while intubating double lumen or nasal endotracheal tube. Conventional video laryngoscope in this study indicates the video laryngoscope blade which has the same curve as Macintosh laryngoscope. It mainly improves the glottic view by front positioning camera.

Anesthesiologist usually place the tip of the blade at vallecula to expose the glottic which is the conventional ways of using Macintosh blade which we name it as Macintosh method. Placing the tip below the epiglottis and lift it up directly is the way of using Miller blade. Theoretically, the Miller method with conventional video laryngoscope may improve the scale of glottic exposure measured with Cormack-Lehane grade. This is a one-group pretest-posttest study to compare the Cormack-Lehane grade with two different methods in the same patient. This study tends to discuss whether this combination can improve the glottic exposure and preserve the advantage of direct laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

1. Aged>20
2. Scheduled to received operation that required general anesthesia with endotracheal tube [3] ASA I, II

Exclusion Criteria:

1. Emergent surgery
2. pregnant
3. Limited mouth opening
4. Poor dental condition
5. Airway obstruction (oral tumor, hypopharyngeal cancer….etc)
6. Deep neck infection
7. Allergic to any anesthetic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Change of cormack lehane grade | Measured from glottic exposed by Macintosh approach to Miller approach. Record the cormack lehane grade. The whole precess will be completed within 5 minutes if there are no difficult intubation.
  Compare the difference of cormack lehane grade using Macintosh ot Miller approach.(cormack lehane grade has four gradings. Grade 1 represent entire glottic opening. Grade 4 represent vocal cord cab not be seen)

SECONDARY OUTCOMES:
Post intubation adverse event | Visit the patient daily at post operation day 1 and record any adverse event until post operation day3 or the patient is discharged.
  Some adverse events are often seen after intubation, such as sore throat, hoarseness....etc.

CONTACTS AND LOCATIONS:
Overall Officials: HAN-LIANG JIANG, MD, Study Chair — Kaohsiung Veterans General Hospital, Department of Anesthesiology
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
We had no experience of making IPD. If it's helpful to other researcher, then we'll try figure out how to do it.

REFERENCES:
- [Background] Serocki G, Bein B, Scholz J, Dorges V. Management of the predicted difficult airway: a comparison of conventional blade laryngoscopy with video-assisted blade laryngoscopy and the GlideScope. Eur J Anaesthesiol. 2010 Jan;27(1):24-30. doi: 10.1097/EJA.0b013e32832d328d. PMID 19809328
- [Background] Kido H, Komasawa N, Matsunami S, Kusaka Y, Minami T. Comparison of McGRATH MAC and Macintosh laryngoscopes for double-lumen endotracheal tube intubation by anesthesia residents: a prospective randomized clinical trial. J Clin Anesth. 2015 Sep;27(6):476-80. doi: 10.1016/j.jclinane.2015.05.011. Epub 2015 Jun 22. PMID 26111665
- [Background] El-Tahan MR, Khidr AM, Gaarour IS, Alshadwi SA, Alghamdi TM, Al'ghamdi A. A Comparison of 3 Videolaryngoscopes for Double-Lumen Tube Intubation in Humans by Users With Mixed Experience: A Randomized Controlled Study. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):277-286. doi: 10.1053/j.jvca.2017.08.009. Epub 2017 Aug 4. PMID 29056498
- [Background] Aziz MF, Abrons RO, Cattano D, Bayman EO, Swanson DE, Hagberg CA, Todd MM, Brambrink AM. First-Attempt Intubation Success of Video Laryngoscopy in Patients with Anticipated Difficult Direct Laryngoscopy: A Multicenter Randomized Controlled Trial Comparing the C-MAC D-Blade Versus the GlideScope in a Mixed Provider and Diverse Patient Population. Anesth Analg. 2016 Mar;122(3):740-750. doi: 10.1213/ANE.0000000000001084. PMID 26579847
- [Background] Liu DX, Ye Y, Zhu YH, Li J, He HY, Dong L, Zhu ZQ. Intubation of non-difficult airways using video laryngoscope versus direct laryngoscope: a randomized, parallel-group study. BMC Anesthesiol. 2019 May 15;19(1):75. doi: 10.1186/s12871-019-0737-3. PMID 31092191
- [Background] Huang P, Zhou R, Lu Z, Hang Y, Wang S, Huang Z. GlideScope(R) versus C-MAC(R)(D) videolaryngoscope versus Macintosh laryngoscope for double lumen endotracheal intubation in patients with predicted normal airways: a randomized, controlled, prospective trial. BMC Anesthesiol. 2020 May 20;20(1):119. doi: 10.1186/s12871-020-01012-y. PMID 32434470

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT05545982/Prot_SAP_000.pdf